CLINICAL TRIAL: NCT03152734
Title: Periinterventional Outcome Study in the Elderly (POSE): European, Multi-centre, Prospective Observational Cohort Study
Brief Title: Periinterventional Outcome Study in the Elderly
Acronym: POSE
Status: Completed | Type: Observational
Sponsor: Mark Coburn (Other)
Responsible Party: Sponsor-Investigator, Mark Coburn, Prof. Dr. med. Mark Coburn, RWTH Aachen University
Organization: RWTH Aachen University (Other)
Other Study IDs: 17-070
Record Dates: First submitted 2017-05-09; First posted 2017-05-15 (Actual); Last update posted 2019-11-20 (Actual); Status verified 2019-11

CONDITIONS: Mortality; Complication, Postoperative
Keywords: Elderly patients, Mortality, morbidity, post-intervention
MeSH Terms: conditions — Postoperative Complications | interventions — Surgical Procedures, Operative

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (1):
- Elderly patient: Elderly patient undergoing surgical and non-surgical intervention with the use of anesthesia provided by an anesthetist
  Interventions: Procedure: Surgical or non-surgical intervention

INTERVENTIONS:
Procedure: Surgical or non-surgical intervention — Each kind of surgical or non-surgical intervention with anesthesia applied by an anesthetist

SUMMARY:
The POSE study will predict critical stages and outcome in a large sample of all surgical and non-surgical interventional patients ≥80 years of age in Europe.

DETAILED DESCRIPTION:
Elderly population (≥80 years) will increase from 5.3% of the total population in 2015 to 9% in 2040. This implies an increasing number and variety of surgical and non-surgical interventional procedures. Little is known about the in-hospital mortality rates in the overall elderly interventional population. Compared with younger interventional patients, the elderly are at greater risk of peri-interventional mortality and morbidity, because of decline in physiological and cognitive reserve, and frequent comorbidities. Previous data are mostly limited to specific populations, like the elderly hip fracture patient.

The investigators aim to recruit as many as possible centers throughout Europe, to participate in this study. A total sample size of 7500 patients will provide reasonable and valid results for the study aims. The primary endpoint will be analysed by fitting a COX-Regression model to the data of the post-interventional mortality until day 30.

ELIGIBILITY:
Inclusion Criteria:

* Age ≥ 80 years
* Written informed consent according to the national law requirements
* All consecutive patients undergoing surgical and non-surgical interventions (e.g. radiological, neuroradiological, cardiological, gastroenterological) with anaesthesia care (done by an anaesthetist) within the selected inclusion period of four weeks
* Elective and emergency procedures
* In-patient and out-patient procedures

Exclusion Criteria:

* People who are institutionalized by court or administrative order
* Patients with re-intervention within the 4 week period, who were already enrolled in this study

Min Age: 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Older Adult
Study Population: Patients will be selected from secondary and tertiary hospitals in several countries in Europe.
Sampling Method: Probability Sample
Enrollment: 9500 (Actual)
Dates: Start 2017-10-01 (Actual); Primary Completion 2019-01-30 (Actual); Study Completion 2019-01-30 (Actual)

PRIMARY OUTCOMES:
Peri-interventional (surgical and non-surgical interventional) all-cause mortality rate on day 30 | From intervention until day 30.
  Number of patients with death from any cause

SECONDARY OUTCOMES:
In-hospital outcome according to the ACS National Surgical Quality Improvement Program® (ACS NSQIP®) | From intervention until day 30.
  Number of patients with e.g. pneumonia, cardiovascular complication, surgical site infection, urinary tract infection, venous thromboembolism, acute or progressive renal failure and re-surgery
Analysis of the new-onset of serious cardiac complications | From intervention up to 30-days after intervention
  Number of patients with serious cardiac complication
  Cardiac complication is defined according to the American Heart Association
Analysis of the new-onset of serious pulmonary complications | From intervention up to 30-days after intervention
  Number of patients with
  * Pneumonia: Clinical or radiological diagnosis. or
  * Pulmonary embolism: Radiological diagnosis. Signs of pneumonia or pulmonary embolism in the autopsy
Analysis of the new-onset of acute stroke | From intervention up to 30-days after intervention
  Number of patients with new-onset of acute stroke, defined as a new focal or generalised neurological deficit of >24h duration in motor, sensory, or coordination functions with compatible brain imaging and confirmed by a neurologist. Transient ischemic attack is not considered as acute stroke. Signs of stroke in the autopsy.
Analysis of the new-onset of acute kidney injury | From intervention up to 30-days after intervention
  Number of patients with new-onset of acute kidney injury, defined according to the AKIN classification as AKI stage ≥2.
  This means increase of creatinine >2-3x from baseline within the hospital stay. Or urine output less than 0.5 ml kg-1 per hour for more than 12 hours. Or signs of acute kidney injury in the autopsy.
Unplanned intensive care unit admission | From intervention until hospital discharge or maximum 30-days after intervention
  Number of patients
Unplanned intubation after intervention | From intervention until hospital discharge or maximum 30-days after intervention
  Number of patients
Hospital discharge destination | From intervention until hospital discharge or maximum 30-days after intervention
  Number of patients, who are not discharged, discharged home, discharged to rehabilitation, discharged to other hospital, discharged to a nursing home, diseased in hospital or discharged to another destination, respectively.
Perioperative admission to a unit with a geriatric care model | From intervention until hospital discharge or maximum 30-days after intervention
  Number of patients, which are post-interventionally admitted to e.g. geriatric units, geriatric co-management models, geriatric liaison services
Patient's functional status of independency | On day 30 after intervention
  Scale assessed by interview of the patient according to the NSQIP (Independent, partially dependent, totally dependent).
Brief screen for cognitive impairment | On day 30 after intervention
  Number of correct recall of three words (Brief Screen for Cognitive Impairment test)
Comparing the postoperative in-hospital and 30-day outcome with preoperatively via NSQIP risk calculator and POSPOM predicted outcome for surgeries | On day 30 after intervention
  Comparing the number of via preoperative NSQIP risk calculator and POSPOM predicted outcomes with the number of postoperative outcomes of the patient
Number of used intra-interventional monitoring for elderly patients in the clinical routine | Intra-interventional
  Number of patients, where a specific monitoring device was intra-interventionally used
Number of patients with premedication | Intra-interventional
  Number of patients with premedication given before intervention.
Type of anesthesia technique | Intra-interventional
  Number of patients with a specific type of anesthesia technique (e.g. spinal, general etc)
Type of the main anesthetic | Intra-interventional
  Number of patients with a specific type of anesthesia drugs (e.g. desflurane, isoflurane etc.)
Type of the main intra-interventional opioid | Intra-interventional
  Number of patients with a specific type of opioid for anesthesia (e.g. fentanyl etc.)
Anesthesia duration | Intra-interventional
  Begin to end of anesthesia for intervention
Amount of intra-interventionally transfused blood and blood products | Intra-interventional
  e.g. transfusion of packed red blood cells, fresh frozen plasmas and platelets
Number of extubated patients | Intra-interventional
  At the end of intervention
Kind of intervention | Intra-interventional
  Surgical procedure category, severity, urgency, wound class
Use of WHO safe surgery checklist | Intra-interventional
  Number of patients , where the WHO safe surgery checklist was used
Kind of referring facility | Pre-interventional at baseline visit
  Number of patients referred from home,other hospital, rehabilitation, nursing home or other referring facility, respectively.
Amount of pre-interventional comorbidities | pre-interventional at baseline visit
  Number of comorbidities
Albumin and hematocrit level before intervention | pre-interventional at baseline visit
  Optional assessment, only if done in the clinical routine
Number of falls in the last 6 months | pre-interventional at baseline visit
  Number of falls per patient
Mini-Cog (for the cognitive status) | pre-interventional at baseline visit
  Performance of the mini-cog test and analysis of the maximum points in this test
Pre-interventional timed "Up & Go" test | pre-interventional at baseline visit
  Seconds to perform the up and go test will be measured
Comparison of the patients' outcomes across Europe | 30 days after intervention
  Comparing the number of adverse outcomes between the hospitals and countries

OTHER OUTCOMES:
Age and gender-effect on the 30 day mortality | 30 days after intervention
  Association of patient age/ gender and mortality
Effect of pre-interventional morbidities on the 30 day mortality | 30 days after intervention
  Association of pre-operative morbidities and mortality
Effect of type of surgery or non-surgical intervention on the 30 day mortality | 30 days after intervention
  Association of type of surgery or non-surgical intervention and mortality
Effect of centre and country on the 30 day mortality | 30 days after intervention
  Association of center/ country and mortality
In-hospital cardiopulmonary resuscitation | From intervention until hospital discharge or maximum 30-days after intervention
  Rate

CONTACTS AND LOCATIONS:
Overall Officials: Mark Coburn, MD, Study Chair — Department of Anesthesiology, University Hospital Aachen, Germany
Locations (177):
- University Hospital Salzburg, Salzburg, Austria
- Belgium (7):
  - ZNA Middelheim, Antwerp
  - Universitair Ziekenhuis Antwerpen, Edegem
  - Ziekenhuis Oost-Limburg, Genk
  - Ghent University Hospital, Ghent
  - AZ Groeninge, Kortrijk
  - University Hospital Leuven, Leuven
  - AZ Turnhout, Turnhout
- Denmark (7):
  - Aarhus Universityhospital, Aarhus
  - Rigshospitalet, Neuroscience Centre, Copenhagen
  - Rigshospitalet, Copenhagen
  - Herlev Hospital, Herlev
  - Nordsjællands Hospital, Hillerød
  - Hospital Unit Horsens, Horsens
  - Hospitaln Lillebælt, Vejle
- France (34):
  - CHU Amiens Picardie, Amiens
  - CHU Angers, Angers
  - Centre Hospitalier Fleyriat, Bourg-en-Bresse
  - Centre hospitalier Pierre Oudot, Bourgoin
  - HIA Clermont Tonnerre, Brest
  - Hopital d'Instruction des Armées Percy, Clamart
  - CH Le Mans, Le Mans
  - Huriez Hospital, University Hospital of Lille, Lille
  - Clinique de la Sauvegarde, Lyon
  - Croix Rousse Hospital, Lyon
  - Hopital Edouard Herriot, Lyon
  - Hôpital Lyon Sud, Lyon
  - Neurologic Hospital-Hospices Civils de Lyon, Lyon
  - AP-HM Hôpital Nord, Marseille
  - CH Martigues, Martigues
  - Clinique Saint Jean, Montpellier
  - Centre Hospitalier Universitaire de Nantes, Nantes
  - CHU Nantes, Nantes
  - AP-HP, Hopital Saint-Louis, Paris
  - Cochin University Hospital, Paris
  - Hopital de la Pitié-Salpe tri ere, Paris
  - Hopital Saint Antoine, Paris
  - Centre Hospitalier Universitaire de Poitiers, Poitiers
  - Hopital Prive Claude Galien, Quincy-sous-Sénart
  - University Hospital of Reims, Reims
  - Clinique Trenel, Saint-Coulomb
  - CHU Hôpital Nord, Saint-Etienne
  - Clinique Mutualiste Saint Etienne, Saint-Etienne
  - Polyclinique de l'atlantique, Saint-Herblain
  - Groupe Hospitalier Selestat-Obernai, Sélestat
  - Hopital Foch, Suresnes
  - Centre Hospitalier de Bigorre, Tarbes
  - CHU Toulouse, Toulouse
  - Gustave Roussy Cancer Center, Villejuif
- Georgia (9):
  - Health centre "Medina", Batumi
  - 5th General Hospital "Open Heart", Tbilisi
  - Acad. N. Kipshidze Central University Clinic, Tbilisi
  - EVEX Traumatology Hospital, Tbilisi
  - Medical Corporation Evex, Tbilisi Referral Hospital, Tbilisi
  - Mediclubgeorgia, Tbilisi
  - New Hospital, Tbilisi
  - Oftalmij, Tbilisi
  - Medical Corporation Evex - Zugdidi Referral Hospital, Zugdidi
- Germany (21):
  - Department of Anesthesiology, University Hospital Aachen, Aachen, North Rhine-Westphalia
  - St. Josef- Hospital, Bochum
  - University Hospital Knappschaftskrankenhaus Bochum, Bochum
  - University of Bonn, Bonn
  - University Hospital Carl Gustav Carus Dresden, Dresden
  - Heinrich-Heine University Duesseldorf, Düsseldorf
  - University Hospital Frankfurt, Frankfurt
  - Hannover Medical School, Hanover
  - Marien Hospital Herne, UK der Ruhr-Universität Bochum, Herne
  - Jena University Hospital, Jena
  - Universitätsklinikum Schleswig-Holstein Campus Luebeck, Lübeck
  - Universitaetsklinikum Marburg, Marburg
  - Johannes Wesling Klinikum Minden, Minden
  - Klinikum der Ludwigs-Maximilians-Universität München (LMU), München
  - Klinikum rechts der Isar der TU München, München
  - St. Franziskus-Hospital Münster, Münster
  - University Hospital Münster, Münster
  - Klinikum Oldenburg AÖR, Oldenburg
  - University Hospital Tübingen, Tübingen
  - Kliniverbund St. Antonius und St. Josef GmbH, Wuppertal
  - University Hospital of Wuerzburg, Würzburg
- Greece (20):
  - Democritus University of Thrace, Alexandroupoli
  - Alexandra Hospital, Athens
  - Evangelismos General Hospital, Athens
  - General Hospital of Athens "G. Gennimatas", Athens
  - Onassis Cardiac Surgery Center, Athens
  - Attikon University Hospital, Chaïdári
  - University Hospital of Ioannina, Ioannina
  - General Hospital of Kavala, Kavala
  - Komotini General Hospital, Komotini
  - University Hospital of Larissa, Larissa
  - University Hospital of Patras, Pátrai
  - Tzaneio General Hospital of Pireaus, Piraeus
  - AHEPA University Hospital, Thessaloniki
  - General Hospital Papanikolaou, Thessaloniki
  - George Papanikolaou, Thessaloniki
  - Hippokrateion General Hospital, Thessaloniki
  - Medical School, Aristotle University of Thessaloniki, Thessaloniki
  - Theagenio Cancer Hospital, Thessaloniki
  - General Hospital of Veroia, Véroia
  - General Hospital of Volos "Achillopouleio", Volos
- Ireland (3):
  - Cork University Hospital Group, Cork
  - St Vincents University Hospital, Dublin
  - Tallaght Hospital, Dublin
- Israel (5):
  - Shaare Zedek Medical Center, Jerusalem
  - Galilee Medical Center, Nahariya
  - Rabin Medical Center Beilinson Hospital, Petah Tikva
  - Sheba Academic Medical Center, Ramat Gan
  - Tel Aviv Sourasky Medical Center, Tel Aviv
- Netherlands (4):
  - Albert Schweitzer Hospital, Dordrecht
  - Maastricht UMC+, Maastricht
  - Maasstad Ziekenhuis, Rotterdam
  - University Medical Center Utrecht, Utrecht
- North Macedonia (2):
  - University Clinic for Gyn & Ob / Clinical Center Mother Teresa, Skopje
  - University Clinic for Traumatology, Orthopedics, Anesthesia, Reanimation, and Intensive Care Medicine, Skopje
- Jagiellonian University Medical College, Krakow, Poland
- Portugal (3):
  - Centro Hospitalar e Universitario de Coimbra, Coimbra
  - Centro Hospitalar Lisboa Norte - Hospital Santa Maria, Lisbon
  - Centro Hospitalar Tamega e Sousa, Penafiel
- Romania (5):
  - Clinical Emergency Hospital of Bucharest, Bucharest
  - Emergency Institute for Cardiovascular Diseases "Prof CC Iliescu", Bucharest
  - Fundeni Clinical Institute, Bucharest
  - University Emergency Central Military Hospital, Bucharest
  - Emergency County Hospital Cluj, Cluj-Napoca
- Russia (4):
  - GBUZ Chelyabinsk Regional Clinical Center of Oncology and Nuclear Medicine, Chelyabinsk
  - Federal State Autonomous Institution N.N. Burdenko National medical research center of neurosurgery of the ministry of health of the Russian federation (N.N. Burdenko NMRCN), Moscow
  - NN Blokhin National Medical Cancer Research Center, Moscow
  - P.A. Herzen Moscow Cancer Research Institute, Moscow
- Serbia (10):
  - Cardiovacular Institute Dedinje, Belgrade
  - CHC Bezaniska Kosa, Belgrade
  - Clinic for ENT and maxillofacial surgery, Clinical Center of Serbia, Belgrade
  - Clinic for orthopedics surgery and traumatology Clinical center of Serbia, Belgrade
  - Clinical Center of Serbia, Cener for anaestesia , Department for digestive surgery, Belgrade
  - Clinical Centre of Serbia, Belgrade
  - Emergency Center, Clinical Center of Serbia, Belgrade
  - Urology Hospital, Clinical center of Serbia, Belgrade
  - Clinical Center Nis, Niš
  - General Hospital Sremska Mitrovica, Sremska Mitrovica
- Spain (17):
  - Hospital Universitario Fundacion Alcorcon, Alcorcón
  - Consorci Sanitari Integral, Barcelona
  - CSI Hospital General de l'Hospitalet, Barcelona
  - Hospital de la Santa Creu i Sant Pau, Barcelona
  - Hospital Universitari Sagrat Cor, Barcelona
  - Universitary General Hospital of Ciudad Real, Ciudad Real
  - Hospital Universitario de Gran Canaria Doctor Negrin, Las Palmas de Gran Canaria
  - Hospital of Leon, León
  - San Pedro Hospital, Logroño
  - Hospital General Gregorio Maranon, Madrid
  - Hospital Ramon y Cajal, Madrid
  - Hospital Universitario Infanta Leonor, Madrid
  - Hospital Universitario La Princesa, Madrid
  - Hospital de Sant Joan Despí Moises Broggi - Consorci Sanitari Integral, Sant Joan Despí
  - Hospital Clinico Universitario, Valencia
  - Hospital Universitario Araba, Vitoria-Gasteiz
  - Hospital Universitario Miguel Servet, Zaragoza
- Switzerland (5):
  - University Hospital Basel, Basel
  - Kantonsspital Baselland Liestal, Liestal
  - Hirslanden Clinic St. Anna Lucern, Lucerne
  - Spital Limmattal, Schlieren
  - Bürgerspital Solothurn, Solothurn
- Turkey (Türkiye) (18):
  - Ankara University Cebeci Hospital, Ankara
  - Ankara University Faculty of Medicine-Ibni Sina Hospital, Ankara
  - Ufuk University Dr. Ridvan Ege Hospital, Ankara
  - University of Health Sciences Diskapi Yildirim Beyazit Education and Training Hospital, Ankara
  - Balikesir Atatürk City Hospital, Balıkesir
  - Kocaeli Derince Training and Research Hospital, Derince
  - TR Ministry of Health Erzurum Palandoken State Hospital, Erzurum
  - Baltalimani Metin Sabanci Bone and Joint Diseases Education and Research Hospital, Istanbul
  - Dr. Siyami Ersek Thoracic and Cardiovascular Surgery Training and Research Hospital, Istanbul
  - Istanbul University, Istanbul Faculty of Medicine, Istanbul
  - Marmara University Pendik Training and Research Hospital, Istanbul
  - Dokuz Eylul University Faculty of Medicine, Izmir
  - Saglik Bilimleri University Tepecik Education and Research Hospital, Izmir
  - Baskent University Konya Research Center, Konya
  - Konya Education and Research Hospital, Konya
  - RTE university school of medicine, Rize
  - Sakarya University School od Medicine, Sakarya
  - Republic of Turkey Ministry of Health Tunceli State Hospital, Tunceli
- Zaporizhzhia State Medical University, Zaporizhzhya, Ukraine

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Hoogma DF, Al Tmimi L, Fieuws S, Tournoy J, Kowark A, Rossaint R, Coburn M, Rex S. Circadian effect of time of anaesthesia on postoperative outcomes in major elective and urgent intervention: a secondary analysis of the Peri-interventional Outcome Study in the Elderly (POSE). Eur J Anaesthesiol Intensive Care. 2022 Aug 24;1(3):e005. doi: 10.1097/EA9.0000000000000005. eCollection 2022 Jun. PMID 39916969
- [Derived] Kowark A, Berger M, Rossaint R, Schmid M, Coburn M; POSE-Study group. Association between benzodiazepine premedication and 30-day mortality rate: A propensity-score weighted analysis of the Peri-interventional Outcome Study in the Elderly (POSE). Eur J Anaesthesiol. 2022 Mar 1;39(3):210-218. doi: 10.1097/EJA.0000000000001638. PMID 34817420
- [Derived] POSE-Study group. Peri-interventional outcome study in the elderly in Europe: A 30-day prospective cohort study. Eur J Anaesthesiol. 2022 Mar 1;39(3):198-209. doi: 10.1097/EJA.0000000000001639. PMID 34799496